CLINICAL TRIAL: NCT05283564
Title: A Pilot Study to Evaluate Percussive Ventilation Breathhold to Improve Lung Stereotactic Ablative Radiotherapy (PVB-SABR)
Brief Title: Study to Evaluate Percussive Ventilation Breathhold to Improve Lung Stereotactic Ablative Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-63842; NCI-2023-00704 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2022-02-24; First posted 2022-03-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Percussive ventilation breathhold (PVB) technique in healthy volunteers (Other): The healthy patient will execute the Percussive ventilation breathhold technique
  Interventions: Other: Percussive Ventilation Breathhold SABR (PVB-SABR)
- Administration of the PVB-SABR in lung cancer patients (Other): Lung cancer patients will execute a PV breathhold and a verification cone-beam CT scan.
  Interventions: Other: Percussive Ventilation Breathhold SABR (PVB-SABR)

INTERVENTIONS:
Other: Percussive Ventilation Breathhold SABR (PVB-SABR) — Number of lung cancer patients with successful administration of PVB technique in PVB-SABR treatment

SUMMARY:
The purpose of this research is to evaluate and determine the rate of successful administration of Percussive ventilation breathhold (PVB) to allow for more accurate radiotherapy for lung tumors.

DETAILED DESCRIPTION:
Primary Objective(s)

* To determine the rate of successful administration of the PVB-SABR in lung cancer patients.
* To determine the rate of successful administration of PVB in healthy volunteers for 5 minutes

Secondary Objective(s)

* To determine the rate of successful administration of PVB in healthy volunteers for 10 minutes as well as for patients' successfully completing the technique for 5 and 10 minutes.
* To collect exploratory clinical (both arms) and dosimetric data from lung cancer patients using PVB-SABR.

ELIGIBILITY:
Inclusion Criteria:

Arm 1: Healthy volunteers age 18 or older

Arm 1: Ability to understand and the willingness to sign (personally or by a legal authorized representative) the written IRB approved informed consent document.

Arm 2: Patients with a diagnosis of primary lung cancer or lung metastases of any primary tumor origin

Arm 2: Patients deemed clinically eligible to be treated with standard of care lung SABR for patient arm

Arm 2: Patients of any gender age 18 or older

Arm 2: Patients with ECOG Performance Status 0-2 and select patients with Performance Status 3 deemed to be suitable candidates based on common sense clinical judgment on the risks versus benefits of SABR

Arm 2: Ability to understand and the willingness to sign (personally or by a legal authorized representative) the written IRB approved informed consent document.

Exclusion Criteria:

Arm 1: No Pregnant Individuals. All individuals of child bearing potential (last menstrual period within the previous 12 months and not surgically sterile) will be tested for pregnancy and documented by study team.

Arm 2: Patients clinically deemed ineligible for standard of care lung SABR treatment for the patient arm (for example, excessive tumor size, individuals who are pregnant or breast feeding, severe pulmonary fibrosis are relative contraindications for lung SABR and are part of standard of care clinical decision making).

Arm 2: Patients with newly-developed pneumothorax

Arm 2: Patients with critical acute illness precluding SABR in the judgment of the treating physician (examples could include active pulmonary embolism and infection requiring inpatient care)

Arm 2: Patients with ECOG Performance Status 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Rate of successful Percussive Ventilation Breathhold (PVB) maneuver in healthy volunteers. | 18 months
  The rate will be measured as the proportion of healthy volunteers who can be successfully execute the Percussive Ventilation Breathhold for 5 minutes. In the event of a failure, both investigator and patient will be asked to specify the reason for failure for purposes of failure analysis.
Rate of successful administration of Percussive Ventilation Breathhold Stereotactic Ablative Radiotherapy (PVB SABR) in lung patients. | 18 months
  The rate will be measured as the proportion of lung cancer patients who successfully complete treatment using the PVB SABR method as defined by 100% of the prescribed Stereotactic Ablative Radiotherapy dose being delivered using the Percussive Ventilation Breathhold (PVB) technique. A failure will be defined as a patient who fails to use the method for any part of the treatment. In the event of a failure, both investigator and patient will be asked to specify the reason for failure for purposes of failure analysis.

SECONDARY OUTCOMES:
Additional time-related endpoints for duration of breathhold with Percussive Ventilation (PV) breathhold intervention for Healthy patients | 3 months
  The rates will be measured as the proportion of healthy volunteers who can be successfully execute the PV breathhold for 10 minutes
Exploratory clinical and dosimetric data on Percussive Ventilation Breathhold Stereotactic Ablative Radiotherapy (PVB SABR) technique | 3 months
  We will collect optional exploratory noninvasive clinical data during PVB including but not limited to real-time CO2 and SpO2 data (using the SenTec Digital Monitoring System or similar device) and surface anatomy monitoring (using devices such as Kinect camera, vision-RT, or laser surface monitoring system). All of these data will be collected on an optional exploratory basis.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson X Mai, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Institute, Palo Alto, California, United States